CLINICAL TRIAL: NCT00696384
Title: An 8-Month Phase 3, Open-Label Study With a Blinded Reversal Phase to Evaluate the Safety and Tolerability of TAK-491 in Subjects With Essential Hypertension
Brief Title: A Safety and Tolerability Study of Azilsartan Medoxomil in Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-491-016; U1111-1113-9088 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2012-01-04 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-11

CONDITIONS: Hypertension
Keywords: Essential Hypertension; Cardiovascular Disease; High Blood Pressure; Drug Therapy
MeSH Terms: conditions — Hypertension; Essential Hypertension; Cardiovascular Diseases | interventions — azilsartan medoxomil; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil QD-Open Label Phase (Baseline - Week 26) (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan Medoxomil QD - Double-Blind Phase (Week 26-32) (Experimental)
  Interventions: Drug: Azilsartan medoxomil, with or without chlorthalidone and other non-angiotensin II receptor blocker antihypertensive medications.
- Placebo QD - Double-Blind Phase (Week 26- 32) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan medoxomil — All subjects initiated azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks, force-titrated to 80 mg, tablets, orally, once daily. After Week 8, chlorthalidone, 25 mg, tablets, orally, once daily as needed and other antihypertensive medications as needed to achieve target blood pressure (defined as <140/90 mm Hg for participants without diabetes or chronic kidney disease (CKD) and <130/80 mm Hg for participants with diabetes or CKD) for up to 26 weeks.
  Study medication could have been up-titrated only after the subject had been at the previous dose level for a minimum of 2 weeks. Study medication could only have been up- or down-titrated by 1 dose level per scheduled or unscheduled visit.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil QD-Open Label Phase (Baseline - Week 26)
Drug: Azilsartan medoxomil, with or without chlorthalidone and other non-angiotensin II receptor blocker antihypertensive medications. — Azilsartan medoxomil at the final dose received during the open-label phase: (20 mg, 40 mg or 80 mg), tablets, orally, once daily with or without chlorthalidone 25 mg, tablets, orally once daily and other non-ARB antihypertensive medications (if currently taking), for 6 weeks/Week 32.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil QD - Double-Blind Phase (Week 26-32)
Drug: Placebo — Azilsartan medoxomil placebo-matching tablets, orally, once daily with or without chlorthalidone 25 mg or other non-ARB antihypertensive (if currently taking), tablets, orally, once daily for 6 weeks/Week 32.
  Arms: Placebo QD - Double-Blind Phase (Week 26- 32)

SUMMARY:
The purpose of this study is to determine the long term safety and tolerability of azilsartan medoxomil, once daily (QD), in participants with Essential Hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure.

A major component of blood pressure regulation is the renin-angiotensin-aldosterone system, a system of hormone-mediated feedback interactions that results in the relaxation or constriction of blood vessels in response to various stimuli. Angiotensin II, a polypeptide hormone, is formed from angiotensin I in a reaction catalyzed by angiotensin-converting enzyme as part of the renin-angiotensin-aldosterone system. AII is the principal pressor agent of the renin-angiotensin-aldosterone system with a myriad of effects on the cardiovascular system and on electrolyte homeostasis. Two receptors for angiotensin II have been identified. Angiotensin II type 1 (AT1) receptors are located predominantly in vascular smooth muscle, where activation by angiotensin II results in vasoconstriction, hypertrophic proliferation, and inflammation. In contrast, stimulation of angiotensin II type 2 (AT2) receptors by angiotensin II results in vasodilation, antiproliferative effects, and other effects that are opposite from those of AT1 receptor stimulation.

Drugs that modulate the renin-angiotensin-aldosterone system are used commonly worldwide for the treatment of hypertension. Of these, some block the synthesis of angiotensin II by inhibiting angiotensin-converting enzyme inhibitors, while others inhibit the action of angiotensin II by binding directly to the AT1 receptor (angiotensin II receptor blockers), thereby allowing blood vessels to dilate, resulting in a reduction in blood pressure. The effects of angiotensin II receptor blockers on other conditions in which the renin-angiotensin-aldosterone system plays a significant role, such as congestive heart failure, post-myocardial infarction management, and diabetic nephropathy, also are being investigated.

Takeda Global Research & Development Center, Inc. is developing TAK-491 (azilsartan medoxomil) to treat mild to moderate essential hypertension. Nonclinical studies have indicated that azilsartan medoxomil is an antagonist of the AT1 receptor subtype.

This study consists of 2 phases. The first phase will be a 26-week, open-label, multicenter phase to evaluate the safety and tolerability of TAK-491 in participants with essential hypertension. Investigators were instructed to manage participants according to a protocol-specified treatment algorithm to achieve target blood pressure. All participants who completed the open-label phase then were randomized into a 6-week double-blind, placebo-controlled (azilsartan medoxomil [maintained at the final dose from the open-label phase] or placebo, in addition to their current other antihypertensive medications including chlorthalidone, as applicable) reversal phase to evaluate maintenance/durability of azilsartan medoxomil -mediated blood pressure reduction, as well as potential rebound following the cessation of azilsartan medoxomil.

Study participation is anticipated to be about 8.5 Months. Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, vital signs including sitting and standing blood pressure and pulse, body height and weight, physical examinations and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria

1. Has essential hypertension (diastolic blood pressure ≥ 95mm Hg and ≤ 119 mm Hg. For participants with diabetes or chronic kidney disease diastolic blood pressure must be ≥ 85 mm Hg and ≤ to 109 mm Hg.
2. Female participant is not of childbearing potential (eg, sterilized, postmenopausal).
3. Female participants of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
4. Clinical laboratory evaluations (including clinical chemistry, hematology, and complete urinalysis) are within the reference range for the testing laboratory unless the results are deemed not clinically significant for inclusion into this study by the investigator.

Exclusion Criteria

1. Systolic blood pressure greater than 185 mm Hg.
2. Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:
3. Is hypersensitive to AII receptor blockers.
4. Recent history (within the last 6 months) of myocardial infarction, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, cerebrovascular accident, or transient ischemic attack.
5. History of moderate to severe heart failure or hypertensive encephalopathy.
6. Has clinically significant cardiac conduction defects (eg, third-degree atrioventricular block, sick sinus syndrome).
7. Has secondary hypertension of any etiology.
8. Known or suspected unilateral or bilateral renal artery stenosis.
9. Has severe renal dysfunction or disease (based on calculated creatinine clearance < 30 mL/min/1.73 m2) at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda
Locations (45):
- United States (33):
  - Huntsville, Alabama
  - Chandler, Arizona
  - Mesa, Arizona
  - Tempe, Arizona
  - Los Gatos, California
  - Sacramento, California
  - Tustin, California
  - Westlake Village, California
  - Colorado Springs, Colorado
  - Wheat Ridge, Colorado
  - Melbourne, Florida
  - Pembroke Pines, Florida
  - Augusta, Georgia
  - South Bend, Indiana
  - Auburn, Maine
  - Marlborough, Massachusetts
  - Chelsea, Michigan
  - St Louis, Missouri
  - Trenton, New Jersey
  - Rochester, New York
  - Burlington, North Carolina
  - Wilmington, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Carlisle, Pennsylvania
  - Philadelphia, Pennsylvania
  - Mt. Pleasant, South Carolina
  - San Antonio, Texas
  - Norfolk, Virginia
  - Lakewood, Washington
  - Renton, Washington
  - Madison, Wisconsin
- Argentina (4):
  - Berazategui, Buenos Aires
  - Pilar, Buenos Aires
  - Córdoba
  - Salta
- Mexico (8):
  - León, Guanajuato
  - Guadalajara, Jalisco
  - Cuernavaca, Morelos
  - Rosario, Santa Fe
  - Tampico, Tamaulipas
  - Durango
  - Mexico City
  - Puebla City

REFERENCES:
- [Derived] Kipnes MS, Handley A, Lloyd E, Barger B, Roberts A. Safety, tolerability, and efficacy of azilsartan medoxomil with or without chlorthalidone during and after 8 months of treatment for hypertension. J Clin Hypertens (Greenwich). 2015 Mar;17(3):183-92. doi: 10.1111/jch.12474. Epub 2015 Jan 24. PMID 25619410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 51 investigative sites in Argentina, Mexico and the United States from 22 June 2007 to 08 May 2009.
Pre-assignment Details: All participants that completed the open-label phase were randomized into a double-blind reversal phase (to continue with azilsartan medoxomil or to placebo, in addition to any other antihypertensive medications received during the open-label phase).
Groups:
- Azilsartan Medoxomil QD - Open Label Phase: All subjects initiated azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks, force-titrated to 80 mg, tablets, orally, once daily. After Week 8, chlorthalidone, 25 mg, tablets, orally, once daily was added as needed, followed by other non-ARB antihypertensive medications as needed to achieve target blood pressure (defined as <140/90 mm Hg for participants without diabetes or chronic kidney disease (CKD) and <130/80 mm Hg for participants with diabetes or CKD) for up to 26 weeks.
  Study medication could have been up-titrated only after the subject had been at the previous dose level for a minimum of 2 weeks. Study medication could only have been up- or down-titrated by 1 dose level per scheduled or unscheduled visit.
- Azilsartan Medoxomil QD - Double-Blind Reversal Phase: Azilsartan medoxomil at the final dose received during the open-label phase: (20 mg, 40 mg or 80 mg), tablets, orally, once daily with or without chlorthalidone 25 mg, tablets, orally once daily and other non-ARB antihypertensive medications (if currently taking), for 6 weeks.
- Placebo QD - Double-Blind Reversal Phase: Azilsartan medoxomil placebo-matching tablets, orally, once daily with or without chlorthalidone 25 mg, orally once daily or other non-ARB antihypertensive (if currently taking), tablets, orally, once daily for 6 weeks.
Period: Open Label Phase
Arm/Group | Azilsartan Medoxomil QD - Open Label Phase | Azilsartan Medoxomil QD - Double-Blind Reversal Phase | Placebo QD - Double-Blind Reversal Phase
Started | 418 | 0 | 0
Completed | 299 | 0 | 0
Not Completed | 119 | 0 | 0
Not completed — Adverse Event | 27 | 0 | 0
Not completed — Protocol Violation | 18 | 0 | 0
Not completed — Lost to Follow-up | 24 | 0 | 0
Not completed — Withdrawal by Subject | 37 | 0 | 0
Not completed — Other | 6 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0
Period: Double Blind Phase
Arm/Group | Azilsartan Medoxomil QD - Open Label Phase | Azilsartan Medoxomil QD - Double-Blind Reversal Phase | Placebo QD - Double-Blind Reversal Phase
Started | 0 | 148 | 151
Completed | 0 | 137 | 145
Not Completed | 0 | 11 | 6
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 3
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Azilsartan Medoxomil QD - Open Label Phase: Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks, titrated to 80 mg, tablets, orally, once daily. After Week 8, chlorthalidone, 25 mg, tablets, orally, once daily as needed and other antihypertensive medications as needed to achieve target blood pressure (defined as <140/90 mm Hg for participants without diabetes or chronic kidney disease (CKD) and <130/80 mm Hg for participants with diabetes or CKD) for up to 26 weeks. Study medication could have been up-titrated only after participant had been at the previous dose level for a minimum of 2 weeks. Study medication could only have been up or down-titrated by 1 dose level per scheduled or unscheduled visit. Baseline characteristics of this Open Label phase population are described in the table below.
Arm/Group | Azilsartan Medoxomil QD - Open Label Phase
Number analyzed (Participants) | 418
Age, Customized [Number; unit: participants]
  <45 years | 89
  Between 45 and 64 years | 287
  ≥ 65 years | 42
Age, Customized [Number; unit: percentage of participants]
  <45 years | 21.3
  Between 45 and 64 years | 68.7
  ≥ 65 years | 10.0
Sex/Gender, Customized [Number; unit: participants]
  Female | 210
  Male | 208

OUTCOME MEASURES:

1. Primary Outcome: Change From Double-blind Baseline (Week 26) in Sitting Clinic Diastolic Blood Pressure to Week 32
Description: The change in sitting clinic diastolic blood pressure measured at final visit or week 32 from Double-blind Baseline/Week 26. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements. Each participant's blood pressure at the Final Visit/Week 26 of the open-label phase represented their Baseline blood pressure for the double-blind reversal phase.
Time Frame: Double-blind Baseline (Week 26) and Week 32.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- Azilsartan Medoxomil QD - Double Blind Reversal Phase: Azilsartan medoxomil at the final dose received during the open-label phase: (20 mg, 40 mg or 80 mg), tablets, orally, once daily with or without chlorthalidone 25 mg, tablets, orally once daily and other non-ARB antihypertensive medications (if currently taking) as needed for 6 weeks.
- Placebo QD - Double Blind Reversal Phase: Azilsartan medoxomil placebo-matching tablets, orally, once daily with or without chlorthalidone 25 mg or other antihypertensive (if currently taking), tablets, orally, once daily for 6 weeks.
Arm/Group | Azilsartan Medoxomil QD - Double Blind Reversal Phase | Placebo QD - Double Blind Reversal Phase
Number analyzed (Participants) | 142 | 148
mmHg | 0.14 (0.726) | 7.92 (0.712)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil QD - Double Blind Reversal Phase vs Placebo QD - Double Blind Reversal Phase; Test type: Superiority or Other; p < 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Includes participants with both a double-blind baseline and postbaseline value; Mean Difference (Final Values) = -7.78, 95% CI 2-sided [-9.78 to -5.78]

2. Secondary Outcome: Change From Double-blind Baseline (Week 26) in Sitting Clinic Systolic Blood Pressure to Week 32
Description: The change in sitting clinic systolic blood pressure measured at final visit or week 32 from Double-blind Baseline/Week 26.. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements. Each participant's blood pressure at the Final Visit/Week 26 of the open-label phase represented their Baseline blood pressure for the double-blind reversal phase.
Time Frame: Double-blind Baseline (Week 26) and Week 32.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil QD - Double Blind Reversal Phase | Placebo QD - Double Blind Reversal Phase
Number analyzed (Participants) | 142 | 148
mmHg | 0.59 (1.121) | 12.97 (1.098)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil QD - Double Blind Reversal Phase vs Placebo QD - Double Blind Reversal Phase; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -12.38, 95% CI 2-sided [-15.47 to -9.29]

3. Secondary Outcome: Change From Open Label Baseline (Week 0) in Sitting Clinic Diastolic Blood Pressure to Week 26
Description: The change from baseline in sitting clinic diastolic blood pressure measured at final visit or week 26.
Time Frame: Baseline and Week 26.
Population: Safety analysis set with last observation carried forward.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil QD - Open Label Phase
Number analyzed (Participants) | 418
mmHg | -15.76 (11.912)

4. Secondary Outcome: Change From Open Label Baseline (Week 0) in Sitting Clinic Systolic Blood Pressure to Week 26
Description: The change from baseline in sitting clinic systolic blood pressure measured at final visit or week 26.
Time Frame: Baseline and Week 26.
Population: Safety analysis set with last observation carried forward.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Azilsartan Medoxomil QD - Open Label Phase
Number analyzed (Participants) | 418
mmHg | -23.01 (20.657)

5. Secondary Outcome: Number of Participants With Adverse Events During the Open-Label Phase
Description: Treatment-emergent adverse events defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after last dose of study drug, or within 30 days after the last dose of study drug for serious adverse event (SAE). A SAE is defined as any untoward medical occurrence that either results in death; is life-threatening; requires hospitalization; results in persistent or significant disability/incapacity; leads to a congenital anomaly/birth defect; or is an important medical event.
Time Frame: Baseline to Week 26
Measure: Number; unit: participants
Groups:
- Azilsartan Medoxomil QD - Open Label Phase: All subjects initiated azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks, force-titrated to 80 mg, tablets, orally, once daily. After Week 8, chlorthalidone, 25 mg, tablets, orally, once daily was added as needed and other non-ARB antihypertensive medications as needed to achieve target blood pressure (defined as <140/90 mm Hg for participants without diabetes or chronic kidney disease (CKD) and <130/80 mm Hg for participants with diabetes or CKD) for up to 26 weeks.
  Study medication could have been up-titrated only after the subject had been at the previous dose level for a minimum of 2 weeks. Study medication could only have been up- or down-titrated by 1 dose level per scheduled or unscheduled visit.
Arm/Group | Azilsartan Medoxomil QD - Open Label Phase
Number analyzed (Participants) | 418
participants
  Serious Adverse Events | 8
  Treatment Emergent Adverse Events | 226

6. Secondary Outcome: Number of Participants With Adverse Events in the Double-Blind Baseline Phase
Description: Treatment-emergent adverse events defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medicinal product reported from first dose of study drug through 14 days after last dose of study drug, or within 30 days after the last dose of study drug for SAE. A SAE is defined as any untoward medical occurrence that either results in death; is life-threatening; requires hospitalization; results in persistent or significant disability/incapacity; leads to a congenital anomaly/birth defect; or is an important medical event.
Time Frame: Double-blind Baseline/Week 26 to Week 32
Measure: Number; unit: participants
Arm/Group | Azilsartan Medoxomil QD - Double Blind Reversal Phase | Placebo QD - Double Blind Reversal Phase
Number analyzed (Participants) | 148 | 151
participants
  Serious Adverse Events | 0 | 1
  Treatment Emergent Adverse Events | 42 | 38

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings.
Groups:
- Azilsartan Medoxomil QD - Open Label: Azilsartan medoxomil 40 mg, tablets, orally, once daily for four weeks, titrated to 80 mg, tablets, orally, once daily.. After Week 8, chlorthalidone, 25 mg, tablets, orally, once daily as needed and other antihypertensive medications as needed to achieve target blood pressure (defined as <140/90 mm Hg for participants without diabetes or chronic kidney disease (CKD) and <130/80 mm Hg for participants with diabetes or CKD) for up to 26 weeks.
  Study medication could have been up-titrated only after the subject had been at the previous dose level for a minimum of 2 weeks. Study medication could only have been up- or down-titrated by 1 dose level per scheduled or unscheduled visit.
- Azilsartan Medoxomil QD - Double-Blind Reversal Phase: Azilsartan medoxomil current dose (20 mg, 40 mg or 80 mg), tablets, orally, once daily with or without chlorthalidone 25 mg, tablets, orally once daily and other antihypertensive medications as needed for 6 weeks.
- Placebo QD - Double-Blind Reversal Phase: Azilsartan medoxomil placebo-matching tablets, orally, once daily with or without chlorthalidone 25 mg or other antihypertensive (if currently taking), tablets, orally, once daily for up to 6 weeks.
Arm/Group | Azilsartan Medoxomil QD - Open Label | Azilsartan Medoxomil QD - Double-Blind Reversal Phase | Placebo QD - Double-Blind Reversal Phase
Serious Adverse Events (participants affected / at risk) | 8/418 | 0/148 | 1/151
Other Adverse Events (participants affected / at risk) | 60/418 | 5/148 | 8/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil QD - Open Label (N=418) | Azilsartan Medoxomil QD - Double-Blind Reversal Phase (N=148) | Placebo QD - Double-Blind Reversal Phase (N=151)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil QD - Open Label (N=418) | Azilsartan Medoxomil QD - Double-Blind Reversal Phase (N=148) | Placebo QD - Double-Blind Reversal Phase (N=151)
Headache (Nervous system disorders) | 30 | 5 | 8
Dizziness (Nervous system disorders) | 36 | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.